CLINICAL TRIAL: NCT03369366
Title: Immediate Reconstruction and Dental Rehabilitation of Maxillofacial Defects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not received.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702812
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Maxillofacial Injuries
Keywords: Maxillofacial Defects; Benign, large tumors requiring surgical resection
MeSH Terms: conditions — Maxillofacial Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reconstruction and Dental Rehabilitation (Experimental): Placement of NobelActive dental implants (minimum of three) using integrated osteotomy and implant placement guide.Placement of provisional screw-retained prosthesis (all while flap is still pedicled to vascular supply). Inset of flap/implant/prosthesis/custom plate construct (KLS Martin Mandibular Reconstruction Implant).
  Interventions: Device: NobelActive; Device: KLS Martin Mandibular Reconstruction Implant

INTERVENTIONS:
Device: NobelActive — NobelActive's expanding tapered implant body condenses bone gradually while the apex with drilling blades enables a smaller osteotomy. These features help to achieve high primary stability in demanding situations, such as soft bone or extraction sockets. NobelActive enables immediate implant placement and Immediate Function where it might otherwise be challenging.
Device: KLS Martin Mandibular Reconstruction Implant — The prefabricated prosthesis will be secured onto the implants using non-engaging multiunit abutments with screws, followed by fixation of the patient-specific plate to the fibula with monocortical screws. The previously used cutting guides are fixated with the screw locations corresponding to the screw locations of the custom plate. This allows for accurate positioning and fixation of the custom construct of the plate and fibula without the need for intermaxillary fixation (IMF).

SUMMARY:
Immediate reconstruction and dental rehabilitation of maxillofacial ablative defects with patient specific reconstruction plates, dental implants, and immediate load provisional screw-retained prosthesis will improve patient short and long term outcomes and improve patient quality of life. Utilizing current technologic advances, patients undergoing large ablative procedures for benign head and neck pathology can now not only have immediate bone and soft tissue reconstruction, but dental rehabilitation as well. Using virtual surgical planning, patient specific selective laser melded reconstruction plates, and dental implants, a screw-retained provisional dental restoration can be fabricated and placed during a one-stage procedure with minimal to no intra-operative prosthetic work required.

DETAILED DESCRIPTION:
The primary goal of any reconstructive procedure is to restore a patient's natural form and function. The new techniques implemented in this study will demonstrate an approach that allows immediate return of the patient's premorbid state in one procedure. The investigators have demonstrated success with a small cohort of patients, and published a recent case study regarding this new technique. This study is meant to build upon the investigators experiences and advance their process and treatment of these patients. With a larger patient population to study, greater data can be obtained, with the ultimate goal of establishing this treatment as a new standard of care for patients with large ablative defects requiring reconstruction.

Patients with benign, large tumors requiring surgical resection with free tissue transfer reconstruction involving the maxilla and mandible will be included in the study. All of the patients will undergo the following pre-operative protocol:

* CT Maxillofacial Region
* CTA
* Dental impression (intra-oral scan and/or impressions)
* Virtual surgical planning
* Patient specific plate fabrication
* Resection and flap harvest osteotomy guides
* Fabrication of screw-retained provisional prosthesis

Surgical treatment protocol involves:

* Resection of benign tumor using osteotomy guides
* Reconstruction with free tissue (osseous free flap) transfer using osteotomy guides
* Placement of dental implants (minimum of three) using integrated osteotomy and implant placement guide
* Placement of provisional screw-retained prosthesis (all while flap is still pedicled to vascular supply)
* Inset of flap/implant/prosthesis/custom plate construct
* Vascular anastomosis and closure

Immediate post-operative management will include a 5-to-7 day post-operative hospital stay and a post-operative CT scan evaluation. Long-term evaluation of patients will include routine clinical exams and cone beam CT scans to evaluate flap and implant survival. Patients, for the purpose of this study, will be followed for one year following placement of final dental prosthesis (18-24 months post-operatively).

ELIGIBILITY:
Inclusion and Exclusion Criteria

Inclusion Criteria:

* Male and Female patients between 16 and 60 years of age
* Patients with benign, large tumors requiring surgical resection with free tissue transfer reconstruction involving the maxilla and mandible will be included in the study.

Exclusion Criteria:

* Patients below the age of 16 years and over the age of 60 years
* Patients with malignant tumors
* Patients with contraindications for surgical intervention and/or free tissue transfer
* Patients actively participating in another investigational clinical study and who, in the Investigator's or opinion, should not be enrolled in this study.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Time to final dental rehabilitation | 6-8 months
  Time elapsed until final dental rehabilitation is reached.

SECONDARY OUTCOMES:
Total operating room time | 6-8 hours
  The total time taken in operating room for a procedure
Surgical outcome accuracy (CT imaging) | 5-10 days post-op
  Accuracy of the proposed surgical outcome assessed via CT scan imaging
Implant survival - Short term | 6 months post operatively
  Six month survival rate of the dental implant
Implant survival - Long term | one year post operatively
  Long term survival rate of the dental implant

CONTACTS AND LOCATIONS:
Overall Officials: Rui P Fernandes, MD, DMD, Principal Investigator — Associate Professor; Associate Chair; Chief, Division of Head and Neck Surgery

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to researchers outside of the study.